CLINICAL TRIAL: NCT01988584
Title: Autologous Cell Therapies for Cerebral Palsy-Chronic (ACT for CP)
Brief Title: Safety and Effectiveness of Banked Cord Blood or Bone Marrow Stem Cells in Children With Cerebral Palsy (CP).
Acronym: ACT for CP
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: The University of Texas Health Science Center, Houston (Other)
Collaborators: Cord Blood Registry, Inc. (Industry); Let's Cure CP Foundation (Other); Mission Connect, a program of TIRR Foundation (Unknown)
Responsible Party: Principal Investigator, Charles Cox, The Children's Fund Distinguished Professor, Department of Pediatric Surgery, The University of Texas Health Science Center, Houston
Allocation: Randomized | Model: Crossover | Masking: Triple | Purpose: Treatment
Other Study IDs: HSC-MS-12-0876
Record Dates: First submitted 2013-11-04; First posted 2013-11-20 (Estimated); Results first posted 2022-11-21 (Actual); Last update posted 2022-11-21 (Actual); Status verified 2022-10

CONDITIONS: Cerebral Palsy
Keywords: Cerebral Palsy; Brain Injury; Stem Cells; Mononuclear Cells; Bone Marrow; Umbilical Cord Blood
MeSH Terms: conditions — Cerebral Palsy; Brain Injuries | interventions — Cell Count

STUDY DESIGN:
Who Masked: Participant, Care Provider, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes

ARMS (4):
- umbilical cord blood (UCB) cells (Experimental): Children who have banked UCB with CBR will receive an umbilical cord blood stem cell infusion at the baseline/treatment visit.
  Interventions: Biological: umbilical cord blood (hUCB) cells
- bone marrow-derived mononuclear cells (BMMNCs) (Experimental): Children in the BMMNC group will undergo bone marrow harvest and stem cell infusion at the baseline/treatment visit.
  Interventions: Biological: bone marrow derived mononuclear cells (BMMNCs)
- saline infusion (placebo), then umbilical cord blood (UCB) cells (Experimental): Five children in each group will be randomly assigned to receive an inactive substance (placebo) at the baseline/treatment visit. Parents will be given the opportunity to cross-over to either the umbilical cord blood or bone marrow harvest group at the one year visit.
  Interventions: Biological: umbilical cord blood (hUCB) cells; Drug: Saline Infusion (Placebo)
- saline infusion (placebo), then bone marrow-derived mononuclear cells (BMMNCs) (Experimental)
  Interventions: Drug: Saline Infusion (Placebo); Biological: bone marrow derived mononuclear cells (BMMNCs)

INTERVENTIONS:
Biological: umbilical cord blood (hUCB) cells — Autologous umbilical cord blood banked with the Cord Blood Registry.
  Other Names: Autolgous Stem Cells
  Arms: saline infusion (placebo), then umbilical cord blood (UCB) cells; umbilical cord blood (UCB) cells
Drug: Saline Infusion (Placebo) — A total of 10 children (5 from each cohort) will be randomized to a placebo infusion at the baseline visit and then have the opportunity to cross-over to stem cell treatment at the 1yr. visit.
  Arms: saline infusion (placebo), then bone marrow-derived mononuclear cells (BMMNCs); saline infusion (placebo), then umbilical cord blood (UCB) cells
Biological: bone marrow derived mononuclear cells (BMMNCs) — Autologous stem cells from bone marrow harvest.
  Other Names: Autologous Stem Cells
  Arms: bone marrow-derived mononuclear cells (BMMNCs); saline infusion (placebo), then bone marrow-derived mononuclear cells (BMMNCs)

SUMMARY:
The purpose of this study is to compare the safety and effectiveness of two types of stem cells,(either banked cord blood or bone marrow), in children between the ages of 2 to 10 years with CP. 15 children with banked cord blood at CBR and 15 children without banked cord blood will be enrolled into the study. The study involves one baseline/treatment visit and 3 follow-up visits at 6 months, 12 months, and 2 years. Five children in each group will be randomized to a placebo control group at the baseline/treatment visit. Parents will not be told if their child received stem cells or a placebo until the 12 month follow-up visit. At that time parents may elect to have their child receive the stem cell treatment; either bone marrow harvest or umbilical cord blood if banked with CBR. All study visits will be conducted at the UTHealth Medical School and Children's Memorial Hermann Hospital in Houston, Texas.

As of 1/21/2014 we have met our enrollment limit for children without banked cord blood undergoing bone marrow harvest for stem cells.

ELIGIBILITY:
Inclusion Criteria:

1. Children with diagnosis of Cerebral Palsy (spastic CP due to periventricular white matter damage or neonatal brain injury from perinatal stroke or intra-ventricular hemorrhage)
2. Gross Motor Function Classification Score level II-V
3. Ages 24 months to 10 years
4. English speaking, if verbal
5. Ability to travel to Houston for treatment and follow-up -

Exclusion Criteria:

1. Known history of:

   * Intractable seizures
   * Traumatic brain injury
   * Genetic disorder (as demonstrated by newborn screening or genetic diagnostic testing)
   * Recently treated or current infection
   * Renal insufficiency or altered renal function (as defined by serum creatinine > 1.5 mg/dl at screening)
   * Hepatic disease or altered liver function (as defined by SGPT > 150 U/L [non-contusion related], and/or T. Bilirubin >1.3 mg/dL at screening)
   * HIV+ (as demonstrated by positive blood test)
   * Immunosuppression (as defined by WBC <3,000 cells/ml at screening)
   * Infectious related neurological injury
   * Sensitivity to Ethylene Oxide (EtO) [found in fumigants and disinfectants]
2. If Athetoid CP diagnosis, other etiologies such as degenerative, mitochondrial, and metabolic disorders must be excluded, and the outcome assessments must be able to be conducted to assess for potential treatment effects
3. Normal brain MRI
4. Evidence of acute illness at the time of infusion, such as, but not limited to, fever (temperature > 37.5 C), vomiting, diarrhea, wheezing or crackles
5. Progressing neurological disease (as defined by Batten Disease, Leukodystrophies, Metabolic disorders, Mitochondrial disorders, Neurotransmitter disorders)
6. Microcephaly, macrocephaly, cortical malformations, genetic disorders of dysgenesis brain malformations due to infection or metabolic disorders
7. Pulmonary disease requiring ventilator support
8. If hUCB candidate, banked cord cells totaling <10 million/kg
9. If hUCB candidate, any positive maternal infectious disease test (Hepatitis A, Hepatitis B, HIV 1, HIV 2, HTLV 1, HTLV 2, and Syphilis)
10. If hUCB candidate, cord blood sample contamination
11. Participation in a concurrent intervention study
12. Unwillingness to return for follow-up visits
13. Contraindications to MRI
14. Any patient that the investigators feel in their opinion the study intervention is unlikely to benefit the patient will be a screen failure.
15. Any patients who are currently or has previously been enrolled in a clinical stem cell study.

Ages: 2 Years to 10 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 20 (Actual)
Dates: Start 2013-11 (Actual); Primary Completion 2018-02-21 (Actual); Study Completion 2018-02-21 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Charles S Cox, MD, Principal Investigator — UTHealth, Medical School, Dept. of Pediatric Surgery
Locations (1):
- UTHealth, Medical School, Dept. of Pediatric Surgery, Houston, Texas, United States

RESULTS

PARTICIPANT FLOW:
Period: Blinded Phase
Arm/Group | Umbilical Cord Blood (UCB) Cells | Bone Marrow-derived Mononuclear Cells (BMMNCs) | Saline Infusion (Placebo), Then Umbilical Cord Blood (UCB) Cells | Saline Infusion (Placebo), Then Bone Marrow-derived Mononuclear Cells (BMMNCs)
Started | 3 | 10 | 2 | 5
12 Month Follow-up | 3 | 9 | 2 | 5
Completed | 3 | 9 | 2 | 4 (One BMMNC Subject Lost To Follow-up After 1yr. Cross-Over Visit)
Not Completed | 0 | 1 | 0 | 1
Period: Unblinded Phase - Placebo Arm Crossover
Arm/Group | Umbilical Cord Blood (UCB) Cells | Bone Marrow-derived Mononuclear Cells (BMMNCs) | Saline Infusion (Placebo), Then Umbilical Cord Blood (UCB) Cells | Saline Infusion (Placebo), Then Bone Marrow-derived Mononuclear Cells (BMMNCs)
Started (Placebo arms cross over to stem cell intervention 12 months after start of study.) | 0 | 0 | 2 | 5
Completed (Crossover arms complete follow-up 12 months after start of stem cell intervention (which is 24 months after start of study).) | 0 | 0 | 2 | 4
Not Completed | 0 | 0 | 0 | 1

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Umbilical Cord Blood (UCB) Cells | Bone Marrow-derived Mononuclear Cells (BMMNCs) | Total
Number analyzed (Participants) | 5 | 15 | 20
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 5 | 15 | 20
  Between 18 and 65 years | 0 | 0 | 0
  >=65 years | 0 | 0 | 0
Age, Continuous [Mean (Standard Deviation); unit: years] | 4 (2.12) | 6.13 (2.92) | 5.6 (2.85)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 2 | 6 | 8
  Male | 3 | 9 | 12
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 1 | 0 | 1
  Not Hispanic or Latino | 4 | 15 | 19
  Unknown or Not Reported | 0 | 0 | 0
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 0 | 0
  Asian | 0 | 2 | 2
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0
  Black or African American | 0 | 0 | 0
  White | 4 | 13 | 17
  More than one race | 1 | 0 | 1
  Unknown or Not Reported | 0 | 0 | 0
Region of Enrollment [Count of Participants; unit: Participants]
  United States | 5 | 13 | 18
  United Kingdom | 0 | 1 | 1
  Italy | 0 | 1 | 1

OUTCOME MEASURES:

1. Primary Outcome: Safety as Assessed by Number of Participants With In-hospital Infusion Toxicity
Description: In-hospital infusion toxicity includes hemodynamic, pulmonary, hepatic, renal, or neurologic complications.
Time Frame: 24 hours after infusion
Measure: Count of Participants; unit: Participants
Groups:
- Saline Infusion (Placebo): saline infusion (placebo): inactive substance
Arm/Group | Umbilical Cord Blood (UCB) Cells | Bone Marrow-derived Mononuclear Cells (BMMNCs) | Saline Infusion (Placebo)
Number analyzed (Participants) | 5 | 15 | 7
Participants | 0 | 0 | 0

2. Primary Outcome: Long-term Safety
Description: Long-term safety as assessed by number of participants who developed new mass lesions or other pathological structural changes or had worsening neurological status
Time Frame: from the time of infusion to 1 year after infusion
Population: Two in the BMMNC arm were lost to follow up.
Measure: Count of Participants; unit: Participants
Arm/Group | Umbilical Cord Blood (UCB) Cells | Bone Marrow-derived Mononuclear Cells (BMMNCs) | Saline Infusion (Placebo)
Number analyzed (Participants) | 5 | 13 | 7
Participants | 0 | 0 | 0

3. Secondary Outcome: Number of Participants With an Improvement in White Matter Integrity.
Description: Number of participants with an improvement in white matter integrity as measured by diffusion tensor imaging (DTI) magnetic resonance imaging (MRI) reconstruction of corticospinal tract (CST) radial diffusivity (RD).
  Improvement is defined as radial diffusivity (RD) decreased in at least one corticospinal tract (CST) reconstruction.
Time Frame: from baseline to 1 year after infusion
Population: Two in the BMMNC arm were lost to follow up.
Measure: Count of Participants; unit: Participants
Arm/Group | Umbilical Cord Blood (UCB) Cells | Bone Marrow-derived Mononuclear Cells (BMMNCs) | Saline Infusion (Placebo)
Number analyzed (Participants) | 5 | 13 | 0
Participants | 5 | 9 | 0

4. Secondary Outcome: Gross Motor Function Classification Score (GMFM-66)
Description: Interval age adjusted scaled scores from 0 to 100 with 0 reflecting a child with low motor ability and 100 indicating high motor ability.
Time Frame: baseline before infusion
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Umbilical Cord Blood (UCB) Cells | Bone Marrow-derived Mononuclear Cells (BMMNCs) | Saline Infusion (Placebo)
Number analyzed (Participants) | 3 | 10 | 7
score on a scale | 43.17 (19.8) | 25.61 (12.83) | 23.24 (15.15)

5. Secondary Outcome: Gross Motor Function Classification Score (GMFM-66)
Description: as for outcome 4
Time Frame: 1 year after infusion
Population: Two in the BMMNC arm were lost to follow up.
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Umbilical Cord Blood (UCB) Cells | Bone Marrow-derived Mononuclear Cells (BMMNCs) | Saline Infusion (Placebo)
Number analyzed (Participants) | 5 | 13 | 0
score on a scale | 36.5 (24.1) | 25.95 (13.88) |

6. Secondary Outcome: Gross Motor Function Classification Score (GMFM-88)
Description: Ordinal age adjusted scaled raw and percent scores from 0 to 100 with 0 reflecting a child with low motor ability and 100 indicating high motor ability.
Time Frame: baseline before infusion
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Umbilical Cord Blood (UCB) Cells | Bone Marrow-derived Mononuclear Cells (BMMNCs) | Saline Infusion (Placebo)
Number analyzed (Participants) | 3 | 10 | 7
score on a scale | 50.67 (37.5) | 24.72 (20.06) | 18.06 (21.56)

7. Secondary Outcome: Gross Motor Function Classification Score (GMFM-88)
Description: as for outcome 6
Time Frame: 1 year after infusion
Population: Two in the BMMNC arm were lost to follow up.
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Umbilical Cord Blood (UCB) Cells | Bone Marrow-derived Mononuclear Cells (BMMNCs) | Saline Infusion (Placebo)
Number analyzed (Participants) | 5 | 13 | 0
score on a scale | 34.77 (40.38) | 25.92 (19.83) |

8. Secondary Outcome: Score on Vineland Adaptive Behavior Scales (VABS-2) - Communication
Description: Standard score ranging from 20 to 140 with higher scores indicate a child with a higher level of functioning and lower scores indicate a lower level of functioning.
Time Frame: baseline before infusion
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Umbilical Cord Blood (UCB) Cells | Bone Marrow-derived Mononuclear Cells (BMMNCs) | Saline Infusion (Placebo)
Number analyzed (Participants) | 3 | 10 | 7
score on a scale | 79 (16.09) | 67.56 (21.04) | 52.86 (15.95)

9. Secondary Outcome: Score on Vineland Adaptive Behavior Scales (VABS-2) - Communication
Description: as for outcome 8
Time Frame: 1 year after infusion
Population: Two in the BMMNC arm were lost to follow up.
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Umbilical Cord Blood (UCB) Cells | Bone Marrow-derived Mononuclear Cells (BMMNCs) | Saline Infusion (Placebo)
Number analyzed (Participants) | 5 | 13 | 0
score on a scale | 64.4 (18.96) | 62.23 (20.79) |

10. Secondary Outcome: Score on Vineland Adaptive Behavior Scales (VABS-2) - Daily Living
Description: as for outcome 8
Time Frame: baseline before infusion
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Umbilical Cord Blood (UCB) Cells | Bone Marrow-derived Mononuclear Cells (BMMNCs) | Saline Infusion (Placebo)
Number analyzed (Participants) | 3 | 10 | 7
score on a scale | 67 (16.09) | 57.44 (9.58) | 49.14 (8.95)

11. Secondary Outcome: Score on Vineland Adaptive Behavior Scales (VABS-2) - Daily Living
Description: as for outcome 8
Time Frame: 1 year after infusion
Population: Two in the BMMNC arm were lost to follow up.
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Umbilical Cord Blood (UCB) Cells | Bone Marrow-derived Mononuclear Cells (BMMNCs) | Saline Infusion (Placebo)
Number analyzed (Participants) | 5 | 13 | 0
score on a scale | 63 (23.16) | 52.54 (13.2) |

12. Secondary Outcome: Score on Vineland Adaptive Behavior Scales (VABS-2) - Social
Description: as for outcome 8
Time Frame: baseline before infusion
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Umbilical Cord Blood (UCB) Cells | Bone Marrow-derived Mononuclear Cells (BMMNCs) | Saline Infusion (Placebo)
Number analyzed (Participants) | 3 | 10 | 7
score on a scale | 83 (13) | 68.89 (19.59) | 57.71 (7.13)

13. Secondary Outcome: Score on Vineland Adaptive Behavior Scales (VABS-2) - Social
Description: as for outcome 8
Time Frame: 1 year after infusion
Population: Two in the BMMNC arm were lost to follow up. One BMMNC subject was untestable at this time point.
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Umbilical Cord Blood (UCB) Cells | Bone Marrow-derived Mononuclear Cells (BMMNCs) | Saline Infusion (Placebo)
Number analyzed (Participants) | 5 | 12 | 0
score on a scale | 65 (16) | 60.75 (16.84) |

14. Secondary Outcome: Score on Vineland Adaptive Behavior Scales (VABS-2) - Motor
Description: as for outcome 8
Time Frame: baseline before infusion
Population: 9 subjects were untestable.
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Umbilical Cord Blood (UCB) Cells | Bone Marrow-derived Mononuclear Cells (BMMNCs) | Saline Infusion (Placebo)
Number analyzed (Participants) | 3 | 4 | 4
score on a scale | 58.67 (15.5) | 43 (11.75) | 38.5 (14.62)

15. Secondary Outcome: Score on Vineland Adaptive Behavior Scales (VABS-2) - Motor
Description: as for outcome 8
Time Frame: 1 year after infusion
Population: Two in the BMMNC arm were lost to follow up. Nine subjects were untestable at this time point.
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Umbilical Cord Blood (UCB) Cells | Bone Marrow-derived Mononuclear Cells (BMMNCs) | Saline Infusion (Placebo)
Number analyzed (Participants) | 3 | 6 | 0
score on a scale | 52.33 (16.8) | 40.67 (11.24) |

16. Secondary Outcome: Score on Pediatric Evaluation of Disability Inventory - Self-Care
Description: Standard scores ranging from 0 to 100 with higher scores indicate a child with a higher level of functioning and lower scores indicate a lower level of functioning.
Time Frame: baseline before infusion
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Umbilical Cord Blood (UCB) Cells | Bone Marrow-derived Mononuclear Cells (BMMNCs) | Saline Infusion (Placebo)
Number analyzed (Participants) | 3 | 10 | 5
score on a scale | 35.4 (12.29) | 43.31 (13.04) | 27.36 (9.35)

17. Secondary Outcome: Score on Pediatric Evaluation of Disability Inventory - Self-Care
Description: as for outcome 16
Time Frame: 1 year after infusion
Population: Two in the BMMNC arm were lost to follow up.
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Umbilical Cord Blood (UCB) Cells | Bone Marrow-derived Mononuclear Cells (BMMNCs) | Saline Infusion (Placebo)
Number analyzed (Participants) | 5 | 13 | 0
score on a scale | 36.28 (13.97) | 37.13 (16.35) |

18. Secondary Outcome: Score on Pediatric Evaluation of Disability Inventory - Mobility
Description: as for outcome 16
Time Frame: baseline before infusion
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Umbilical Cord Blood (UCB) Cells | Bone Marrow-derived Mononuclear Cells (BMMNCs) | Saline Infusion (Placebo)
Number analyzed (Participants) | 3 | 10 | 5
score on a scale | 46.83 (27.62) | 33.31 (11.91) | 26.54 (12.88)

19. Secondary Outcome: Score on Pediatric Evaluation of Disability Inventory - Mobility
Description: as for outcome 16
Time Frame: 1 year after infusion
Population: Two in the BMMNC arm were lost to follow up.
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Umbilical Cord Blood (UCB) Cells | Bone Marrow-derived Mononuclear Cells (BMMNCs) | Saline Infusion (Placebo)
Number analyzed (Participants) | 5 | 13 | 0
score on a scale | 39.66 (36.36) | 34.16 (14.8) |

20. Secondary Outcome: Score on Pediatric Evaluation of Disability Inventory - Social
Description: as for outcome 16
Time Frame: baseline before infusion
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Umbilical Cord Blood (UCB) Cells | Bone Marrow-derived Mononuclear Cells (BMMNCs) | Saline Infusion (Placebo)
Number analyzed (Participants) | 3 | 10 | 5
score on a scale | 46.9 (7.82) | 52 (12.02) | 34.12 (16.15)

21. Secondary Outcome: Score on Pediatric Evaluation of Disability Inventory - Social
Description: as for outcome 16
Time Frame: 1 year after infusion
Population: Two in the BMMNC arm were lost to follow up.
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Umbilical Cord Blood (UCB) Cells | Bone Marrow-derived Mononuclear Cells (BMMNCs) | Saline Infusion (Placebo)
Number analyzed (Participants) | 5 | 13 | 0
score on a scale | 44.54 (9.29) | 47.32 (14.82) |

22. Secondary Outcome: Score on A Developmental NEuroPSYchological Assessment (NEPSY-II) - Learning and Memory Memory Subtest - Recall
Description: Scales scores from 1 to 19 with higher scores indicate better outcomes and lower scores indicate poorer outcomes.
Time Frame: baseline before infusion
Population: Data were not collected for the 5 in the UCB cell arm and 4 in the placebo arm. Untestable with this instrument.
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Umbilical Cord Blood (UCB) Cells | Bone Marrow-derived Mononuclear Cells (BMMNCs) | Saline Infusion (Placebo)
Number analyzed (Participants) | 0 | 10 | 1
score on a scale |  | 8.33 (0.58) | 6 (0)

23. Secondary Outcome: Score on A Developmental NEuroPSYchological Assessment (NEPSY-II) - Learning and Memory Memory Subtest - Recall
Description: Scales scores from 1 to 19 with higher scores indicate better outcomes and lower scores indicate poorer outcomes.
Time Frame: 1 year after infusion
Population: Only 4 subjects were testable at this time point.
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Umbilical Cord Blood (UCB) Cells | Bone Marrow-derived Mononuclear Cells (BMMNCs) | Saline Infusion (Placebo)
Number analyzed (Participants) | 1 | 3 | 0
score on a scale | 6 (0) | 5 (1) |

24. Secondary Outcome: Score on A Developmental NEuroPSYchological Assessment (NEPSY-II) - Learning and Memory Memory Subtest - Free/Cued
Description: Scales scores from 1 to 19 with higher scores indicate better outcomes and lower scores indicate poorer outcomes.
Time Frame: baseline before infusion
Population: Only 4 subjects were testable at this time point.
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Umbilical Cord Blood (UCB) Cells | Bone Marrow-derived Mononuclear Cells (BMMNCs) | Saline Infusion (Placebo)
Number analyzed (Participants) | 0 | 3 | 1
score on a scale |  | 5.67 (1.53) | 6 (0)

25. Secondary Outcome: Score on A Developmental NEuroPSYchological Assessment (NEPSY-II) - Learning and Memory Memory Subtest - Free/Cued
Description: Scales scores from 1 to 19 with higher scores indicate better outcomes and lower scores indicate poorer outcomes.
Time Frame: 1 year after infusion
Population: Only 3 subjects were testable at this time point.
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Umbilical Cord Blood (UCB) Cells | Bone Marrow-derived Mononuclear Cells (BMMNCs) | Saline Infusion (Placebo)
Number analyzed (Participants) | 0 | 3 | 0
score on a scale |  | 4 (0) |

26. Secondary Outcome: Expressive and Receptive Vocabulary as Assessed by Score on the Peabody Picture Vocabulary Test (PPVT-4)
Description: Standard score ranging from 20 to 160. Higher scores indicate a child with a higher level of functioning and lower scores indicate a lower level of functioning.
Time Frame: baseline before infusion
Population: Only 7 subjects were testable with this instrument.
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Umbilical Cord Blood (UCB) Cells | Bone Marrow-derived Mononuclear Cells (BMMNCs) | Saline Infusion (Placebo)
Number analyzed (Participants) | 2 | 4 | 1
score on a scale | 80 (26.87) | 85 (13.34) | 89 (0)

27. Secondary Outcome: Expressive and Receptive Vocabulary as Assessed by Score on the Peabody Picture Vocabulary Test (PPVT-4)
Description: as for outcome 26
Time Frame: 1 year after infusion
Population: Only 6 subjects were testable at this time point.
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Umbilical Cord Blood (UCB) Cells | Bone Marrow-derived Mononuclear Cells (BMMNCs) | Saline Infusion (Placebo)
Number analyzed (Participants) | 2 | 4 | 0
score on a scale | 56.5 (21.92) | 86 (11.58) |

28. Secondary Outcome: Score on Cerebral Palsy Quality of Life Questionnaire (CPQOL) - Family
Description: as for outcome 16
Time Frame: baseline before infusion
Population: Only 7 subjects were testable with this instrument.
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Umbilical Cord Blood (UCB) Cells | Bone Marrow-derived Mononuclear Cells (BMMNCs) | Saline Infusion (Placebo)
Number analyzed (Participants) | 1 | 4 | 2
score on a scale | 87.5 (0) | 75.78 (15.39) | 75 (36.36)

29. Secondary Outcome: Score on Cerebral Palsy Quality of Life Questionnaire (CPQOL) - Family
Description: as for outcome 16
Time Frame: 1 year after infusion
Population: Two in the BMMNC arm were lost to follow up.
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Umbilical Cord Blood (UCB) Cells | Bone Marrow-derived Mononuclear Cells (BMMNCs) | Saline Infusion (Placebo)
Number analyzed (Participants) | 4 | 10 | 0
score on a scale | 79.69 (22.89) | 72.81 (17.74) |

30. Secondary Outcome: Score on Cerebral Palsy Quality of Life Questionnaire (CPQOL) - Social
Description: as for outcome 16
Time Frame: baseline before infusion
Population: Only 8 subjects were testable with this instrument
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Umbilical Cord Blood (UCB) Cells | Bone Marrow-derived Mononuclear Cells (BMMNCs) | Saline Infusion (Placebo)
Number analyzed (Participants) | 1 | 4 | 3
score on a scale | 88.64 (0) | 75.57 (9.75) | 83.71 (15.01)

31. Secondary Outcome: Score on Cerebral Palsy Quality of Life Questionnaire (CPQOL) - Social
Description: as for outcome 16
Time Frame: 1 year after infusion
Population: Two in the BMMNC arm were lost to follow up. Five subjects were untestable.
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Umbilical Cord Blood (UCB) Cells | Bone Marrow-derived Mononuclear Cells (BMMNCs) | Saline Infusion (Placebo)
Number analyzed (Participants) | 4 | 10 | 0
score on a scale | 87.7 (8.67) | 74.77 (9.21) |

32. Secondary Outcome: Score on Cerebral Palsy Quality of Life Questionnaire (CPQOL) - Feelings
Description: as for outcome 16
Time Frame: baseline before infusion
Population: 13 subjects were testable with this instrument.
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Umbilical Cord Blood (UCB) Cells | Bone Marrow-derived Mononuclear Cells (BMMNCs) | Saline Infusion (Placebo)
Number analyzed (Participants) | 0 | 10 | 3
score on a scale |  | 60.16 (6.1) | 48.96 (2.76)

33. Secondary Outcome: Score on Cerebral Palsy Quality of Life Questionnaire (CPQOL) - Feelings
Description: as for outcome 16
Time Frame: 1 year after infusion
Population: Two in the BMMNC arm were lost to follow up. Five subjects were untestable.
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Umbilical Cord Blood (UCB) Cells | Bone Marrow-derived Mononuclear Cells (BMMNCs) | Saline Infusion (Placebo)
Number analyzed (Participants) | 3 | 10 | 0
score on a scale | 67.01 (26.85) | 55.73 (9.68) |

34. Secondary Outcome: Score on Cerebral Palsy Quality of Life Questionnaire (CPQOL) - Participation
Description: as for outcome 16
Time Frame: baseline before infusion
Population: Only 8 subjects were testable with this instrument.
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Umbilical Cord Blood (UCB) Cells | Bone Marrow-derived Mononuclear Cells (BMMNCs) | Saline Infusion (Placebo)
Number analyzed (Participants) | 1 | 4 | 3
score on a scale | 72.73 (0) | 56.82 (8.25) | 56.82 (17.71)

35. Secondary Outcome: Score on Cerebral Palsy Quality of Life Questionnaire (CPQOL) - Participation
Description: as for outcome 16
Time Frame: 1 year after infusion
Population: Two in the BMMNC arm were lost to follow up. Five subjects were untestable at this time point.
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Umbilical Cord Blood (UCB) Cells | Bone Marrow-derived Mononuclear Cells (BMMNCs) | Saline Infusion (Placebo)
Number analyzed (Participants) | 4 | 9 | 0
score on a scale | 69.88 (18.57) | 55.81 (8.74) |

36. Secondary Outcome: Score on Cerebral Palsy Quality of Life Questionnaire (CPQOL) - Emotional
Description: as for outcome 16
Time Frame: baseline before infusion
Population: Only 8 subjects were testable with this instrument.
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Umbilical Cord Blood (UCB) Cells | Bone Marrow-derived Mononuclear Cells (BMMNCs) | Saline Infusion (Placebo)
Number analyzed (Participants) | 1 | 4 | 3
score on a scale | 85.42 (0) | 75.52 (5.98) | 69.44 (6.7)

37. Secondary Outcome: Score on Cerebral Palsy Quality of Life Questionnaire (CPQOL) - Emotional
Description: as for outcome 16
Time Frame: 1 year after infusion
Population: Two in the BMMNC arm were lost to follow up. Five other subjects were untestable at this time point.
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Umbilical Cord Blood (UCB) Cells | Bone Marrow-derived Mononuclear Cells (BMMNCs) | Saline Infusion (Placebo)
Number analyzed (Participants) | 4 | 10 | 0
score on a scale | 78.12 (15.73) | 70.83 (8.56) |

38. Secondary Outcome: Score on Cerebral Palsy Quality of Life Questionnaire (CPQOL) - Access
Description: as for outcome 16
Time Frame: baseline before infusion
Population: Only 8 subjects were testable with this instrument.
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Umbilical Cord Blood (UCB) Cells | Bone Marrow-derived Mononuclear Cells (BMMNCs) | Saline Infusion (Placebo)
Number analyzed (Participants) | 1 | 4 | 3
score on a scale | 47.5 (0) | 63.75 (10.31) | 80.83 (17.02)

39. Secondary Outcome: Score on Cerebral Palsy Quality of Life Questionnaire (CPQOL) - Access
Description: as for outcome 16
Time Frame: 1 year after infusion
Population: Two in the BMMNC arm were lost to follow up. Five subjects were untestable at this time point.
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Umbilical Cord Blood (UCB) Cells | Bone Marrow-derived Mononuclear Cells (BMMNCs) | Saline Infusion (Placebo)
Number analyzed (Participants) | 4 | 10 | 0
score on a scale | 72.5 (29.01) | 65.5 (10.26) |

40. Secondary Outcome: Score on Cerebral Palsy Quality of Life Questionnaire (CPQOL) - Pain
Description: as for outcome 16
Time Frame: baseline before infusion
Population: Only 7 subjects were testable with this instrument.
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Umbilical Cord Blood (UCB) Cells | Bone Marrow-derived Mononuclear Cells (BMMNCs) | Saline Infusion (Placebo)
Number analyzed (Participants) | 1 | 4 | 2
score on a scale | 3.13 (0) | 40.63 (20.53) | 35.94 (19.88)

41. Secondary Outcome: Score on Cerebral Palsy Quality of Life Questionnaire (CPQOL) - Pain
Description: as for outcome 16
Time Frame: 1 year after infusion
Population: Two in the BMMNC arm were lost to follow up. Eight subjects were untestable at this time point.
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Umbilical Cord Blood (UCB) Cells | Bone Marrow-derived Mononuclear Cells (BMMNCs) | Saline Infusion (Placebo)
Number analyzed (Participants) | 2 | 9 | 0
score on a scale | 22.39 (20.82) | 34.38 (21.26) |

42. Secondary Outcome: Visual-Spatial Processing as Assessed by Score on the Motor-Free Visual Perception Test (MVPT-3)
Description: Standard scores ranging from 55 to 145 with higher scores indicating better outcomes and lower scores poorer outcomes.
Time Frame: baseline before infusion
Population: Only three subjects were testable with this instrument.
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Umbilical Cord Blood (UCB) Cells | Bone Marrow-derived Mononuclear Cells (BMMNCs) | Saline Infusion (Placebo)
Number analyzed (Participants) | 1 | 2 | 0
score on a scale | 55 (0) | 55 (0) |

43. Secondary Outcome: Visual-Spatial Processing as Assessed by Score on the Motor-Free Visual Perception Test (MVPT-3)
Description: Standard scores ranging from 55 to 145 with higher scores indicating better outcomes and lower scores poorer outcomes.
Time Frame: 1 year after infusion
Population: Data were not collected for the 5 in the UCB cell arm.
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Umbilical Cord Blood (UCB) Cells | Bone Marrow-derived Mononuclear Cells (BMMNCs) | Saline Infusion (Placebo)
Number analyzed (Participants) | 0 | 2 | 0
score on a scale |  | 63 (11.31) |

ADVERSE EVENTS:
Time Frame: 1 year
Description: Serious Adverse Events (SAEs) were defined using the the Common Terminology Criteria for Adverse Events (CTCAE) V5.0. All SAEs and AEs are reported, and all SAEs and AEs were deemed to be unrelated to the stem cell intervention.
Arm/Group | Umbilical Cord Blood (UCB) Cells | Bone Marrow-derived Mononuclear Cells (BMMNCs) | Saline Infusion (Placebo)
All-Cause Mortality (participants affected / at risk) | 0/5 | 0/15 | 0/7
Serious Adverse Events (participants affected / at risk) | 2/5 | 3/15 | 0/7
Other Adverse Events (participants affected / at risk) | 1/5 | 8/15 | 3/7
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Umbilical Cord Blood (UCB) Cells (N=5) | Bone Marrow-derived Mononuclear Cells (BMMNCs) (N=15) | Saline Infusion (Placebo) (N=7)
Upper Tract Respiratory Infection (Infections and infestations) | 0 (0) | 2 (2) | 0 (0)
Febrile Convulsion (Febrile Seizure) (Nervous system disorders) | 1 (1) | 0 (0) | 0 (0)
Osteotomy (Planned Hip Osteotomy) (Surgical and medical procedures) | 1 (1) | 0 (0) | 0 (0)
Pneumonia (Infections and infestations) | 0 (0) | 1 (1) | 0 (0)
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Umbilical Cord Blood (UCB) Cells (N=5) | Bone Marrow-derived Mononuclear Cells (BMMNCs) (N=15) | Saline Infusion (Placebo) (N=7)
Epistaxis (Nose Bleed) (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 0 (0) | 1 (1)
Gastroenteritis (Stomach Flu) (Infections and infestations) | 0 (0) | 2 (3) | 0 (0)
Ear Infection (Infections and infestations) | 0 (0) | 2 (2) | 0 (0)
Seizures (More Frequent Seizures) (Nervous system disorders) | 1 (1) | 1 (1) | 1 (1)
Vitiligo (Skin and subcutaneous tissue disorders) | 0 (0) | 1 (1) | 0 (0)
Haematochezia (Bloody Stools/Chrohn's Disease) (Gastrointestinal disorders) | 0 (0) | 0 (0) | 1 (1)
Nasal Congestion (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 1 (1) | 0 (0)
Pneumonia (Infections and infestations) | 1 (1) | 0 (0) | 0 (0)
Croup Infectious (Infections and infestations) | 1 (1) | 0 (0) | 0 (0)
Upper Respiratory Tract Infection (Infections and infestations) | 1 (1) | 2 (2) | 0 (0)
Respiratory Tract Infection (Infections and infestations) | 0 (0) | 0 (0) | 1 (2)

LIMITATIONS AND CAVEATS:
Limitations common to treating heterogeneous conditions and to cell based therapies. First, patients enrolled had wide range of clinical and imaging findings, which made pooling small data sample problematic. Imaging studies are problematic with hemispheric volume loss secondary to in utero stroke, etc. Second, variability in available cord blood doses. Due to a competing trial, few US families with banked autologous units and not already treated. Unable to reach target enrollment.

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2017-10-23): https://cdn.clinicaltrials.gov/large-docs/84/NCT01988584/Prot_SAP_000.pdf